CLINICAL TRIAL: NCT04070079
Title: Evaluation of Intrahepatic Immune and Virological Response to Tenofovir Alafenamide With Fine Needle Aspiration Biopsy in Chronic Hepatitis B: an Investigator-Initiated, Cohort Study
Brief Title: Tenofovir Alafenamide With Fine Needle Aspiration Biopsy in Chronic Hepatitis B:
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Harry Janssen, Chief of Hepatology | Director Toronto Centre for Liver Disease | Director Viral Hepatitis Care Network (VIRCAN) | Professor of Medicine, University of Toronto |, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-US-320-4667
Record Dates: First submitted 2019-03-29; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tenofovir Alafenamide (Other): Tenofovir Alafenamide 25mg, Dosed orally, once daily with or without food.
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — TAF 25mg once daily orally, for 48 weeks

SUMMARY:
The objective of this study is to identify immunological mechanisms that contribute to normalization of liver inflammation in chronic hepatitis B (CHB) patients starting the antiviral nucleoside analogue, Tenofovir alafenamide (TAF).

DETAILED DESCRIPTION:
Investigator-initiated, phase 4 study in which recruited patients will receive, TAF 25mg once daily, for 48 weeks (Figure 1 and Table 1). The total duration of the study to End of Follow-up (EOF) will be 48 weeks. After Week 48, participants will be offered 2 years of TAF therapy. Sample collection 0, 12, 24 w was chosen to analyze immune responses based on ALT normalization rates. This mono-center study will be conducted at Toronto Centre for Liver Disease, Canada.

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 years

  * Chronic hepatitis B (HBsAg positive ≥ six months)
  * HBeAg positive or negative
  * ALT >19 for females and >30 for males (AASLD criteria)
  * HBV DNA>4 log IU/mL for HBeAg positive and >3 log for HBeAg negative patients
  * No oral antiviral treatment or IFN for ≥6 months
  * Adequate contraception. For males, at least one method of contraception should be used and for females, a barrier contraception method should be used in combination with one other form of contraception.
  * Written informed consent

Exclusion Criteria:

* • Treatment with any investigational drug within 60 days of entry into this protocol

  * Immune-suppressive treatment within the previous 6 months
  * History of decompensated cirrhosis (defined as direct (conjugated)
  * bilirubin > 1.2 × ULN,
  * prothrombin time (PT) > 1.2 × ULN
  * platelets < 100,000/mm3
  * serum albumin < 3.5 g/dL
  * prior history of clinical hepatic decompensation (jaundice in the presence of cirrhosis, ascites, gastric bleeding, oesophageal varices or encephalopathy)
  * Liver transplantation
  * Co-infection with hepatitis C virus, hepatitis D virus or HIV
  * Other significant liver disease: alcoholic liver disease, drug-related liver disease, auto-immune hepatitis, hemochromatosis, Wilson's disease or alpha-1 antitrypsin deficiency
  * Estimated glomerular filtration rate <50 mL/min/1.73m2 or any significant renal disease.
  * Alpha-fetoprotein > 50 ng/ml
  * Pregnancy, breast-feeding
  * Other significant medical illness that might interfere with this study: significant pulmonary dysfunction in previous 6 months, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g. HIV positivity, auto-immune diseases, organ transplants other than cornea and hair transplant)
  * Substance abuse, such as alcohol (≥80 g/day), I.V. drugs and inhaled drugs in past 2 years. Current methadone usage is allowed.
  * Any other condition which in the opinion of the investigator would make the patient unsuitable for enrolment, or could interfere with the patient participating in and completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
TAF-mediated reduction of inflammatory gene expression in intraheaptic immune cells | 3 years
  Longitudinal samples collected from each patient will be used to measure changes in intrahepatic and peripheral innate and adaptive immune composition, function and gene expression from baseline to ALT normalization after starting TAF.
TAF-mediated reduction of serological markers of HBV replication | 3 years
  Existing and experimental biomarkers of HBV replication will be measured to compare the viral response to the immune response
  1. HBsAg/HBeAg seroclearance
  2. HBsAg/HBeAg seroconversion,
  3. Serum quantitative HBsAg/HBeAg levels,
  4. Serum HBV DNA levels
  5. HBV RNA levels
  6. Hepatitis B core-related Antigen (HBcrAg) levels;
  7. ALT levels.
TAF-mediated reduction of intrahepatic HBV replication intermediates and cccDNA levels | 3 years
  HBV replication intermediates and cccDNA measured as copies/mg of liver tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided yet.